CLINICAL TRIAL: NCT00004106
Title: Phase II Trial of Temozolomide for the Treatment of Mycosis Fungoides and the Sezary Syndrome
Brief Title: Temozolomide in Treating Patients With Mycosis Fungoides or Sezary Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per Data Monitoring Committee given the poor/inadequate accrual.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU FDA97H3; NU-FDA97H3; NCI-G99-1597; STU00010001 (Other: Northwestern University IRB)
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide — Temozolomid will be administered orally at a dose of 150mg/m2/day for 5 days for a total of 4 weeks

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying temozolomide to see how well it works in treating patients with mycosis fungoides or Sezary syndrome that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate to temozolomide in patients with relapsed mycosis fungoides or Sezary syndrome.
* Determine the toxic effects of this drug in these patients.
* Correlate pretreatment AGT activity in tumor cells with response to this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral temozolomide once daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity for a maximum of 1 year.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mycosis fungoides or Sezary syndrome

  * Stage IB-IVB disease
  * Must have failed at least one prior systemic therapy
  * Generalized erythroderma allowed
* Measurable disease and at least one indicator lesion OR evaluable disease for erythrodermic patients only

  * Prior radiotherapy to areas of measurable disease allowed if disease progression is present in the site or if measurable disease is present outside irradiation port

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.2 mg/dL
* SGOT or SGPT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No clinically significant peripheral venous insufficiency

Other:

* HIV negative
* No poorly controlled diabetes mellitus
* No acute infection requiring IV antibiotics
* No other medical condition that would prevent ingestion or absorption of oral medication
* No other neoplasm within the past 5 years except curatively treated squamous cell or basal cell skin cancer, melanoma in situ, or carcinoma in situ of the cervix
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior biologic therapy and recovered
* No concurrent growth factors or epoetin alfa

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* At least 4 weeks since prior topical steroids

Radiotherapy:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy for local control or palliation and recovered

Surgery:

* Recovered from prior major surgery

Other:

* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 1998-05; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Response rate | After every 2 cycles of therapy
  Disease response will be assessed using bi-dimensional measurements of lesions with clearly defined margins by medical photograph (skin lesion) or by radiological imaging (internal lesions).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (3):
- United States (3):
  - Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois